CLINICAL TRIAL: NCT00359892
Title: A Multi-Center, Open-Label Phase II Study of Single-Agent GX15-070MS Administered as a 24-Hour Infusion Every 2 Weeks to Patients With Relapsed or Refractory Hodgkin's Lymphoma
Brief Title: Safety and Efficacy of Obatoclax Mesylate (GX15-070MS) in the Treatment of Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gemin X (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEM011
Record Dates: First submitted 2006-08-02; First posted 2006-08-03 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Hodgkin's Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — obatoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Obatoclax Mesylate (Experimental): Obatoclax Mesylate 60mg
  Interventions: Drug: Obatoclax mesylate (GX15-070MS)

INTERVENTIONS:
Drug: Obatoclax mesylate (GX15-070MS) — 60 mg q2wks

SUMMARY:
Defects in the apoptotic process can lead to the onset of cancer by allowing cells to grow unchecked when an oncogenic signal is present. Obatoclax is designed to restore apoptosis through inhibition of the Bcl-2 family of proteins, thereby reinstating the natural process of cell death that is often inhibited in cancer cells.

This is a multi-center, open-label, Phase II study of single-agent obatoclax administered in 2-week cycles as a 24-hour infusion every 2 weeks at a fixed dose of 60 mg to patients with relapsed or refractory Hodgkin's Lymphoma. Infusions may be administered on an out-patient basis. No investigational or commercial agents or therapies other than those described in the protocol may be administered with the intent to treat the patient's malignancy. Supportive care measures including those directed at controlling symptoms resulting from Hodgkin's Lymphoma (blood products, growth factor, etc.) are allowed.

ELIGIBILITY:
Inclusion Criteria:

* Pathological confirmation of Hodgkin's Lymphoma.
* Must have measurable disease.
* Evidence of progressive disease following at least one prior line of combination therapy.
* Must have failed, refused, or otherwise not a candidate for stem cell transplant.
* Patient's must have normal organ function.
* Willing to submit to blood sampling for planned PK and PD analyses.
* Ability to understand and willingness to sign a written informed consent form.

Exclusion Criteria:

* No other agents or therapies administered with the intent to treat malignancy.
* Patients with prior exposure to obatoclax.
* Prior allogeneic stem cell transplant if evidence of graft versus host disease, or requirement for steroids or other immunosuppressive therapy.
* Uncontrolled, intercurrent illness.
* Pregnant women and women who are breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-07; Primary Completion 2007-09 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Determine the response rate to obatoclax and characterize the safety profile; Determine the steady-state pharmacokinetic parameters and pharmacodynamic response. | 4 weeks to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jean Viallet, MD, Study Director — Gemin X, Inc.
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Oki Y, Copeland A, Hagemeister F, Fayad LE, Fanale M, Romaguera J, Younes A. Experience with obatoclax mesylate (GX15-070), a small molecule pan-Bcl-2 family antagonist in patients with relapsed or refractory classical Hodgkin lymphoma. Blood. 2012 Mar 1;119(9):2171-2. doi: 10.1182/blood-2011-11-391037. No abstract available. PMID 22383790